CLINICAL TRIAL: NCT06579469
Title: Prospective Evaluation Of Delayed Effects Of Pediatric Car T Cell Therapy (PROSPER)
Brief Title: Prospective Evaluation Of Delayed Effects Of Pediatric Car T Cell Therapy
Status: Recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Rally Foundation for Childhood Cancer Research (Other)
Responsible Party: Sponsor
Other Study IDs: PROSPER; NCI-2024-06836 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2024-08-28; First posted 2024-08-30 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: B-ALL; Hematologic Malignancy; Solid Tumor
Keywords: CAR T cell infusion; Late Effects
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and bone marrow
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- B cell acute lymphoblastic leukemia (B cell acute lymphoblastic leukemia (B-ALL) ) cohort: B-ALL participants who have received initial CAR T cell therapy within the last 1-3 months.
- Other hematologic malignancy: Other hematologic malignancy participants who have received initial CAR T cell therapy within the last 1-3 months.
- Solid tumor (ST): ST participants who have received initial CAR T cell therapy within the last 1-3 months.

SUMMARY:
This study is being done to learn more about the short-term and long-term side effects of CAR-T cell therapy. Specifically, researchers want to know how often patients get infections, have delays in recovering blood cell counts and/or have damage to the nervous system.

DETAILED DESCRIPTION:
Primary Objectives

* Bone Marrow Function: To report on the incidence, timing, severity of, and risk factors for bone marrow dysfunction in participants in remission or without bone marrow involvement of disease at 3- and 6-months following CAR T cell therapy. (B-ALL cohort)
* Infection/Immune Reconstitution: To evaluate the incidence, timing, severity of and risk factors for clinically significant infections following CAR T cell therapy at 3- and 6-months following CAR T cell therapy. (B-ALL cohort)
* Neurotoxicity: To evaluate the incidence, timing, severity of, and risk factors for persistent ICANS at 3- and 6-months post CAR T cell therapy. (B-ALL cohort)

Secondary Objectives

* To evaluate bone marrow function, infection/immune reconstitution, and neurotoxicity at 12 months and 24 months post CAR T cell therapy in participants with B-ALL.
* To characterize bone marrow function, infection/immune reconstitution, and neurotoxicity between 3 and 24 months after CAR T cell therapy in other hematologic malignancies and solid tumor cohorts.

Participants will have an assessment of preexisting morbidity and potential risk factors, collection of specimens for banking, scheduled late effects monitoring, laboratory analysis, and screening studies. Data and biospecimens will be collected at 3 months, 6 months, 1 year and 2 years after CAR T cell infusion.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have received an initial systemically-administered CAR T cell infusion within the last 1-3 months (+/- 14 days).

  * Initial infusion is defined as the first administration of a CAR T cell product the participant has not previously received OR receipt of a CAR T cell product previously received after an interval allogeneic HSCT.
* Age ≤ 30 years at CAR T cell infusion.

Exclusion Criteria:

* Active malignancy other than the disease under study.
* Planned consolidative HSCT within 3 months post CAR T cell infusion.
* Received or planned additional disease directed therapy post CAR T cell infusion.
* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants who have received CAR T cell therapy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-20 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Presence of bone marrow dysfunction (BMD) | Within 6 months post CAR T-cell therapy
  Among patients in remission or without bone marrow involvement of disease in the B-ALL cohort, we will summarize the rates of prevalent BMD at 3- and 6-months post-infusion and estimate the cumulative incidence of new BMD and BMD recovery for patients with prevalent BMD at 3- and 6-months.
Occurrence of clinically significant infections | Within 6 months post CAR T-cell therapy
  The infection density of clinically significant infections in 3-6 months will be summarized in the B-ALL cohort.
Presence of persistent ICANS | Within 6 months post CAR T-cell therapy
  We will summarize the rates of persistent ICANS at 3- and 6-months post-infusion and estimate the cumulative incidence and timing of new ICANS and ICANS recovery for patients with persistent ICANS at 3- and 6-months in the B-ALL cohort.

SECONDARY OUTCOMES:
Presence of bone marrow dysfunction (BMD) | Within 24 months post CAR T-cell therapy
  Among patients in remission or without bone marrow involvement of disease in the B-ALL cohort, we will summarize the rates of prevalent BMD at 12- and 24-months post-infusion and estimate the cumulative incidence of new BMD and BMD recovery for patients with prevalent BMD at 12- and 24-months. Analyses will be replicated in the other hematologic malignancies and solid tumor cohorts.
Severity of BMD | Within 24 months post CAR T-cell therapy
  The highest severity BMD for each patient will be recorded. The severity of BMD in the B-ALL cohort will be described using descriptive statistics. Analyses will be replicated in the other hematologic malignancies and solid tumor cohorts.
Occurrence of clinically significant infections | Within 24 months post CAR T-cell therapy
  The infection density of clinically significant infections within 24 months will be summarized in the B-ALL cohort. Analyses will be replicated in the other hematologic malignancies and solid tumor cohorts.
Time to the earliest clinically significant infection | Within 24 months post CAR T-cell therapy
  The time from 3 months post-infusion to the first clinically significant post-infusion within 24 months post-infusion will be summarized in the B-ALL cohort. The cumulative incidence of the first clinically significant infection post-infusion within 24 months will be estimated in B-ALL cohort. Analyses will be replicated in the other hematologic malignancies and solid tumor cohorts.
Severity of clinically significant infections | Within 24 months post CAR T-cell therapy
  The highest severity among all clinically significant infections for each patient will be summarized. The severity of clinically significant infections in the B-ALL cohort will be described. Analyses will be replicated in the other hematologic malignancies and solid tumor cohorts.
Presence of persistent ICANS | Within 24 months post CAR T-cell therapy
  We will summarize the rates of persistent ICANS at 12- and 24-months post-infusion and estimate the cumulative incidence and timing of new ICANS and ICANS recovery for patients with persistent ICANS at 12- and 24-months in B-ALL cohort. Analyses will be replicated in the other hematologic malignancies and solid tumor cohorts.
Severity of persistent ICANS | Within 24 months post CAR T-cell therapy
  The highest severity of ICANS for each patient will be recorded. The severity of ICANS in the B-ALL cohort will be described using descriptive statistics. Analyses will be replicated in the other hematologic malignancies and solid tumor cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Epperly, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (2):
- United States (2):
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Children's Hospital of Wisconsin., Milwaukee, Wisconsin

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols